CLINICAL TRIAL: NCT06426550
Title: Clinical and Microbiological Evaluation of Laser Therapy in the Treatment of Periodontal Disease in Stages III and IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriela Alessandra da Cruz Galhardo Camargo, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 78007624.4.0000.5626
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Periodontitis; Periodontitis, Adult
Keywords: Periodontal Diseases; Periodontal Pocket; Laser Therapy; Methylene Blue
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis; Periodontal Diseases; Periodontal Pocket | interventions — Periodontal Index

STUDY DESIGN:
Intervention Model Description: Clinical, laboratory, longitudinal split-mouth study carried out in humans.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by a blind clinician for the initial assessment of participants, using a computer program (Spyder 5.5.4), in which each patient will be randomly selected to define the site to receive one of the treatments. Next, gels will be encoded in a syringe and applied by a researcher blind to the sites and reagents, each of the 4 sites will receive one of the following treatments: 1 - photosensitization with 0.005% AM gel (Fórmula e Ação Farmácia, São Paulo, SP, Brazil) for 5 minutes, and apply photodynamic therapy with a red laser; 2 - photobiomodulation with red laser; 3 - photobiomodulation with infrared laser; and 4 - control, application of saline gel and, after 5 minutes, simulate the application of the laser, with the device in inactive mode, in order to maintain blinding of the patients (control). In groups 2 and 3, as no gel will be applied, the application of the gel with an empty syringe will be simulated, to keep patients blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Photodynamic therapy and 0.005% methylene blue (PDT) (Experimental): Photosensitization will be performed with 0.005% methylene blue gel for 5 minutes, and photodynamic therapy will be applied with a red laser (660 nm) using a DuoⓇ laser with the optical fiber inside the periodontal pocket in back and forth movements, for 90s, 9 joules of energy, dose of 508.5J/cm2, irradiance of 5.65W/cm2 and power of 100mW.
  Interventions: Procedure: Periodontal treatment
- Photobiomodulation with a red laser (PBMV) (Experimental): Photobiomodulation will be performed with a red laser (660 nm) using a DuoⓇ laser with the optical fiber inside the periodontal pocket in back and forth movements, for 90s, 9 joules of energy, dose of 508.5J/cm2, irradiance of 5.65W/cm2 and power of 100mW. The application of the gel with an empty syringe will be simulated, and waited 5 minutes.
  Interventions: Procedure: Periodontal treatment
- Photobiomodulation with an infrared laser (PBMIV) (Experimental): Photobiomodulation will be performed with an infrared laser (808 nm) using a DuoⓇ laser with the optical fiber inside the periodontal pocket in back and forth movements, for 90s, 9 joules of energy, dose of 508.5J/cm2, irradiance of 5.65W/cm2 and power of 100mW. The application of the gel with an empty syringe will be simulated, and waited 5 minutes.
  Interventions: Procedure: Periodontal treatment
- Saline solution - Control (C) (Placebo Comparator): Saline gel will be applied in the periodontal pocket and, after 5 minutes, the laser application will be simulated, with the device in inactive mode.
  Interventions: Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: Periodontal treatment — Conventional periodontal treatment, scaling and root planning, will be performed with ultrasound (Dabi Atlante, Rio de Janeiro, RJ, Brazil) complemented with Gracey curettes (Golgran, São Caetano do Sul, SP, Brazil) on each patient under local anesthesia. The maintenance therapy will include professional plaque control and scaling and root planning in recurrent periodontal pockets, every 30 days, until 3 months, when the periodontal parameters will be reassessed.

SUMMARY:
The aim of this clinical trial is to evaluate photodynamic therapy and photobiomodulation in the periodontitis treatment. To evaluate the clinical and microbiological response of conventional periodontal treatment associated with photodynamic therapy and photobiomodulation with red or infrared laser.

Participants will receive periodontal treatment carried out with the use 0.005% methylene blue and laser therapy (photodynamic therapy), associated with conventional periodontal treatment, as well as the use of photobiomodulation with red or infrared laser associated with conventional periodontal treatment in participants with periodontitis. So, twenty periodontitis patients will be selected and separated in two groups compared with placebo. Clinical and microbiological parameters will be evaluated at baseline and 3 months after periodontal treatment: plaque Index, bleeding on probe, probing depth, gingival recession and clinical attachment level.

DETAILED DESCRIPTION:
Periodontitis is a chronic, inflammatory and multifactorial disease, caused by an interaction between debiotic biofilm and its products and an exacerbated host response, leading to the progressive destruction of the supporting periodontium (bone, cement and periodontal ligament), causing loss of clinical attachment. and radiographic, bleeding on probing and periodontal pocket formation. Periodontal disease has a high prevalence and is one of the main causes of edentulism, with a great negative impact on chewing function, aesthetics and quality of life related to oral health. It is, therefore, considered a serious public health problem.

Conventional periodontal therapy consists of scaling and root planing (SRP) and control of supragingival plaque, but in some cases it has been shown to be ineffective in treating periodontitis, especially in difficult to access areas such as furcations and deep pockets. These cases benefit from adjuvant therapies, such as laser therapy, to help heal periodontal tissues, reduce microorganisms and improve clinical parameters.

Photobiomodulation and photodynamic therapy have been widely applied in the treatment of periodontal disease, due to their clinical, cellular and bactericidal effects. When associated with conventional periodontal therapy, its benefits increase, promoting a significant reduction in probing depth, number of deep pockets and bleeding. Furthermore, significant reduction of periodontopathogens and Candida albicans can be observed in the literature after photobiomodulation and photodynamic therapy.

Despite the benefits found when different laser therapy protocols are used in periodontal treatment, due to the lack of studies with high methodological quality and weak evidence in the existing literature, more studies are needed to prove their effects, establish appropriate protocols and evaluate the antimicrobial potential in periodontopathogens, which remains debatable, as recent systematic reviews point out.

The direct benefits of this study are the treatment of periodontal disease for the participants and for the scientific community to indicate new forms of periodontal therapy using different protocols of laser therapy associated with periodontal instrumentation. All tooth pocket sites in all groups will receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with periodontal disease;
* Four or more periodontal sites with PPD≥6 mm and CAL≥5 mm, non-adjacent;
* Generalized periodontitis, with more than 30% of the sites involved (Caton et al., 2018);
* Stages III and IV of periodontal disease (Caton et al., 2018);

Exclusion Criteria:

* Participants with hypersensitivity to the components of the 0.005% methylene blue gel;
* Received periodontal treatment in the last six months;
* Drugs (alcoholics, use of anti-inflammatories and antibiotics in the last 3 months);

Any evidence of systemic modifying factors which may directly interfere with the completion of the work (bias), such as:

* Pregnant and breastfeeding women;
* Hormone replacement therapy;
* Smoking;
* Hyperglycemia;
* Osteoporosis;
* Diagnosed with HIV+ or AIDS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Plaque index (PI) | Baseline and 3 months
  Plaque index will be expressed in percentage per individual to evaluate the supragingival plaque control.
Bleeding on probing (BOP) | Baseline and 3 months
  Bleeding on probing (BOP) will be expressed in percentage per individual to evaluate presence of BOP <20% good results.
Pocket probing depth (PPD) | Baseline and 3 months
  Pocket probing depth (PPD) will be evaluated in millimeters. The measure will be performed at six sites per tooth using a periodontal probe. The PPD corresponds to the distance from the gingival margin to the apical portion of the gingival sulcus or periodontal pocket.
Gingival recession (GR) | Baseline and 3 months
  Gingival recession (GR) will be measured clinically in millimeters with a periodontal probe as the distance from the cemento-enamel junction to the depth of the free gingival margin.
Clinical attachment level (CAL) | Baseline and 3 months
  Clinical attachment level (CAL) will be measured clinically in millimeters with a periodontal probe and corresponds as the distance from the cemento-enamel junction to the base of the periodontal pocket. CAL represents the extension of periodontal support that has been lost around a tooth.

SECONDARY OUTCOMES:
Microbiogical analysis | Baseline and 3 months
  Pooled biofilms from gingival fluid of four sites with PPD with 6 mm or more will be collected to evaluate the presence of periodontal pathogens. The samples will be collected from the selected sites and stored in eppendorfs with PBS 1X in -20oC until the microbiological analyses, that will consist in DNA extraction, electroforesis and qualitative polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela AC Camargo, Doctor, Principal Investigator — Fluminense Federal University
Locations (1):
- Fluminense Federal University, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
The result will be communicated verbally to each participant.

REFERENCES:
- [Background] Akram Z, Al-Shareef SA, Daood U, Asiri FY, Shah AH, AlQahtani MA, Vohra F, Javed F. Bactericidal Efficacy of Photodynamic Therapy Against Periodontal Pathogens in Periodontal Disease: A Systematic Review. Photomed Laser Surg. 2016 Apr;34(4):137-49. doi: 10.1089/pho.2015.4076. Epub 2016 Mar 16. PMID 26982216
- [Background] Akram Z. How effective is adjunctive antimicrobial photodynamic therapy in treating deep periodontal pockets in periodontal disease? A systematic review. J Investig Clin Dent. 2018 Nov;9(4):e12345. doi: 10.1111/jicd.12345. Epub 2018 Jun 4. PMID 29863310
- [Background] Ren C, McGrath C, Jin L, Zhang C, Yang Y. The effectiveness of low-level laser therapy as an adjunct to non-surgical periodontal treatment: a meta-analysis. J Periodontal Res. 2017 Feb;52(1):8-20. doi: 10.1111/jre.12361. Epub 2016 Mar 2. PMID 26932392